CLINICAL TRIAL: NCT02313233
Title: Research on Benefit of Umooze as Add-on Therapy in Benign Prostatic Hyperplasia
Brief Title: Research on Benefit of Umooze as Add- on Therapy in Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRC01110908
Record Dates: First submitted 2014-12-05; First posted 2014-12-10 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umooze (Experimental): Tablet oral dosage. Astragalus radix Extracts 480 mg+ Soy extracts 20 mg
  Interventions: Dietary Supplement: Umooze
- Placebo (Placebo Comparator): Cornstarch.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Umooze — Umooze is consisted of Astragalus radix extracts and soy extracts. Astragalus radix (AR) is the dried root of Astragalus membranaceus Bge. Var. mongholicus and is used as a tonic in the traditional Chinese medicine. According to the reports submitted by the National Cancer institute of American, people who eat soybean products can reduce the incidence rate for prostate cancer. The composition of Umooze is invented by Golden Biotechnology Corp. against prostatic hyperplasia.
  Arms: Umooze
Dietary Supplement: Placebo — Placebo is consisted of cornstarch and is provided by by Golden Biotechnology Corp.
  Arms: Placebo

SUMMARY:
To evaluate the improvement in symptoms of Benign Prostatic Hyperplasia (BPH) according to the Prostate Symptom Score (IPSS) and Quality- of- Life (QoL) index after add- on therapy of Umooze twice daily administration for 56 days in patients with BPH.

DETAILED DESCRIPTION:
The study product, Umooze, contain Astragalus radix extracts and Soy extracts as the combination of 960:40 in one 500 mg tablet. Umooze is sold in the market as food. The objective of this study is to evaluate the benefit of Umooze as add- on therapy in BPH, by evaluation the improvement in symptoms of BPH assessed according to the International Prostate Symptom Score (IPSS) and Quality- of- Life (QoL) index after add- on therapy of Umooze in patients with BPH. The IPSS is a validated 7-item urinary symptom severity scale.

A randomized, two-regimen, placebo-controlled, parallel- design is used in this study in which each subject will receive Umooze or placebo. The add- on study product will be administered twice daily for 56 days. Benefit will be evaluated at baseline and subsequently on the study day 28, 42, and 56, such as IPSS index, QoL index, Qmax, PVR, prostate volume and Prostate-specific antigen(PSA).

ELIGIBILITY:
Inclusion Criteria:

* Males aged >=40 years old
* Screened by inquiry and diagnosed as BPH based on the result of a digital rectal examination (DRE) or transrectal ultrasonography (TRUS)
* Prostate volume >= 20 cm3
* Has complained of voiding symptoms related to BPH
* Has an IPSS >= 13 or an UFR measure of Qmax <= 15 ml/sec together with a voided volume >= 150 ml.
* Serum PSA < 6.5 ng/ml
* Has been treated with medication for BPH
* Informed consent form signed.

Exclusion Criteria:

* Sensitivity to study product
* Had received prostatic surgery for BPH during the past 24 weeks
* Hard nodule found by DRE
* Ongoing neurogenic bladder, urinary tract infection, bladder stone, urethral stricture, bladder cancer, prostate cancer, severe liver dysfunction, severe renal dysfunction or severe cardiovascular disease.
* Patient has clinically significant physical disability or abnormal findings on physical examination or laboratory testing judged by the investigator or co- investigator.
* Participation of any clinical investigation during the last 30 days.
* Individuals are judged by the investigators or co- investigator to be undesirable as subjects.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ching- Chia Li, M.D, Principal Investigator — Kaohsiung Municipal Ta-Tung Hospital
Locations (1):
- Kaohsiung Municipal TA- TUNG Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angalakuditi M, Seifert RF, Hayes RP, O'Leary MP, Viktrup L. Measurement properties of the benign prostatic hyperplasia impact index in tadalafil studies. Health Qual Life Outcomes. 2010 Nov 12;8:131. doi: 10.1186/1477-7525-8-131. PMID 21073697
- [Background] Li NC, Chen S, Yang XH, Du LD, Wang JY, Na YQ; Beijing Tamsulosin Study Group. Efficacy of low-dose tamsulosin in chinese patients with symptomatic benign prostatic hyperplasia. Clin Drug Investig. 2003;23(12):781-7. doi: 10.2165/00044011-200323120-00003. PMID 17536892
- [Background] Upadhyay L, Tripathi K, Kulkarni KS. A study of prostane in the treatment of benign prostatic hyperplasia. Phytother Res. 2001 Aug;15(5):411-5. doi: 10.1002/ptr.769. PMID 11507733
- [Background] Gaynor ML. Isoflavones and the prevention and treatment of prostate disease: is there a role? Cleve Clin J Med. 2003 Mar;70(3):203-4, 206, 208-9 passim. doi: 10.3949/ccjm.70.3.203. PMID 12678210
- [Background] Kurashige S, Akuzawa Y, Endo F. Effects of astragali radix extract on carcinogenesis, cytokine production, and cytotoxicity in mice treated with a carcinogen, N-butyl-N'-butanolnitrosoamine. Cancer Invest. 1999;17(1):30-5. doi: 10.1080/07357909909011714. PMID 10999046
- [Background] Lin J, Dong HF, Oppenheim JJ, Howard OM. Effects of astragali radix on the growth of different cancer cell lines. World J Gastroenterol. 2003 Apr;9(4):670-3. doi: 10.3748/wjg.v9.i4.670. PMID 12679907
- [Background] Messina M, Redmond G. Effects of soy protein and soybean isoflavones on thyroid function in healthy adults and hypothyroid patients: a review of the relevant literature. Thyroid. 2006 Mar;16(3):249-58. doi: 10.1089/thy.2006.16.249. PMID 16571087
- [Background] Safety, efficacy and impact on Patients' quality of life of a long-term treatment with the alpha(1)-blocker alfuzosin in symptomatic patients with BPH. The Italian Alfuzosin Co-Operative Group. Eur Urol. 2000 Jun;37(6):680-6. doi: 10.1159/000020218. PMID 10828668

RESULTS

PARTICIPANT FLOW:
Groups:
- Umooze: Tablet oral dosage. Astragalus radix Extracts 480 mg+ Soy extract 20 mg
  Umooze: Umooze is consisted of Astragalus radix extracts and soy isoflavones. Astragalus radix (AR) is the dried root of Astragalus membranaceus Bge. Var. mongholicus and is used as a tonic in the traditional Chinese medicine. According to the reports submitted by the National Cancer institute of American, people who eat soybean products can reduce the incidence rate for prostate cancer. The composition of Umooze is invented by Golden Biotechnology Corp. against prostatic hyperplasia. Umooze is given as add-on therapy for benigh prostate hyperplasia (BPH). All the subjects have the history for this medical condition and receive the medication. Each subject receives Umooze in the morning and evening for a continuous 56- day. Each oral dose of Umooze was given 2 tablets with about 240 ml of water.
- Placebo: Cornstarch is used as placebo. It's taken for the subjects who are diagnosed as benign prostate hyperplasia (BPH) and given medication only once a day before going to bed. Each subject receives the placebo in the morning and evening for a continuous 56- day. Each oral dose of placebo was given 2 tablets with about 240 ml of water.
Period: Overall Study
Arm/Group | Umooze | Placebo
Started | 20 | 21
Completed | 18 | 18
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Administrative reason | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis includes the International Prostate Symptom Score (IPSS), quality-of-life (QoL), urinary flow rate (Qmax), postvoided residual volume (PVR), prostate volume, serum PSA level. All the subjects have the history of benigh prostate hyperplasia and have been receiving the medication for this condition.
Groups:
- Umooze: Tablet oral dosage. Astragalus radix Extracts 480 mg+ Soy extract 20 mg
  Umooze: Umooze is consisted of Astragalus radix extracts and soy isoflavones. Astragalus radix (AR) is the dried root of Astragalus membranaceus Bge. Var. mongholicus and is used as a tonic in the traditional Chinese medicine. According to the reports submitted by the National Cancer institute of American, people who eat soybean products can reduce the incidence rate for prostate cancer. The composition of Umooze is invented by Golden Biotechnology Corp. against prostatic hyperplasia. The study product is given as add- on therapy in BPH. All the eligible subjects included in this study have the history for benign prostate hyperplasia (BPH) and receive the medication for this condition. Each subject receives the Umooze in the morning and evening for a continuous 56- day. Each oral dose of Umooze was given 2 tablets with about 240 ml of water.
- Total: Total of all reporting groups
Arm/Group | Umooze | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 7 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 18 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 18 | 18 | 36
Internation Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — The international prostate symptom score (IPSS) is a validated 7- item urinary symptom severity scale. The answers are assigned from 0 to 5, indicating increasing severity. The total score therefore ranges from 0 to 35 points (asymptomatic to symptomatic). Patients can be classified as follows: <=7 is mildly symptomatic; 8~ 19 is moderately symptomatic; 20~ 35 is severely symptomatic.
  units on a scale | 13.22 (6.26) | 19.5 (8.03) | 16.36 (7.67)
Quality-of-Life [Mean (Standard Deviation); unit: units on a scale] — The QoL index is a single question with scores of 0-6 point and corresponding to the assessment index ranging from delighted to terrible.
  units on a scale | 3.33 (1.50) | 3.78 (1.22) | 3.56 (1.34)
Uroflowmetry (UFR) measure of maximum flow rate (Qmax) [Mean (Standard Deviation); unit: ml/ sec] — Urine flow rate is a measure of the quantity of urine excreted. Qmax is an indicator to diagnose the enlarged prostate. A lower Qmax may relate to the pressure on the urethra by the enlarged prostate.
  ml/ sec | 11.5 (2.88) | 10.23 (3.71) | 10.85 (3.29)
Postvoid Residual Volume (PVR) [Mean (Standard Deviation); unit: ml] — This PVR test measures the quantity of urine remained in the bladder after urination. This test is helpful to evaluate the existence of urination problems including an enlarged prostate (BPH).
  ml | 43.7 (27.6) | 52.4 (67.0) | 48.06 (50.00)
Prostate volume [Mean (Standard Deviation); unit: cm^3] — The measurement of prostate volume is used to diagnose an abnormal enlargement of the prostate. Abnormally enlarged prostate may be caused by inflammation or viral infection.
  cm^3 | 37.2 (20.1) | 39.5 (16.9) | 39.10 (18.51)
Serum Total Prostate-Specific Antigen level (PSA) [Mean (Standard Deviation); unit: nanograms/ ml] — The prostate- specific antigen (PSA) is a protein produced by the prostate gland. This test is utilized to evaluate the presence of prostate hyperplasia if a rise of PSA level detected in a man's blood.
  nanograms/ ml | 1.54 (1.34) | 1.95 (1.31) | 1.74 (1.31)
Different original medications and dosages [Number; unit: participants] — The study product (Umooze or placebo) is given as add-on therapy in BPH, therefore the evaluation of benefit may be affected by the original medication.
  participants
    Harnalidge® 0.4 mg QD treatment | 11 | 11 | 22
    Harnalidge® 0.2 mg QD treatment | 2 | 3 | 5
    Harnalidge® 0.1 mg QD treatment | 1 | 0 | 1
    Doxaben® 4 mg QD treatment | 2 | 2 | 4
    Doxaben® XL 4 mg QD treatment | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS)
Description: It's 7- item urinary symptom severity scale. The answers are assigned points from 0 to 5, indicating increasing severity. The total score can therefore range from 0 to 35 points.
Time Frame: 56 days
Population: For all subjects' medical histories in this study, there are one subject receiving Hatnalidge 0.1 mg once daily (QD), five subjects receiving Harnalidge 0.2 mg QD, 22 subjects receiving Harnalidge 0.4 mg QD and eight subjects receiving Doxaben 4 mg or Doxaben XL 4 mg QD for BPH treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Umooze: Tablet oral dosage. Astragalus radix Extracts 480 mg+ Soy bean Extracts 20 mg
  Umooze: Umooze is consisted of Astragalus radix extracts and soy isoflavones. Astragalus radix (AR) is the dried root of Astragalus membranaceus Bge. Var. mongholicus and is used as a tonic in the traditional Chinese medicine. According to the reports submitted by the National Cancer institute of American, people who eat soybean products can reduce the incidence rate for prostate cancer. The composition of Umooze is invented by Golden Biotechnology Corp. against prostatic hyperplasia. Umooze is used as add- on therapy for the subjects who take the medication for benign prostate hyperplasia (BPH). Each subject receives the study product in the morning and evening for a continuous 56- day. Each oral dose of Umooze was given 2 tablets with about 240 ml of water.
- Placebo: Cornstarch is used as placebo. Each subject receives the placebo in the morning and evening for a continuous 56- day. Each oral dose of placebo was given 2 tablets with about 240 ml of water.
Arm/Group | Umooze | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  International prostate symptom score | 9.83 (4.48) | 13.6 (6.88)
  Difference in IPSS between V1 and V6 | -3.39 (6.11) | -5.94 (8.11)

2. Secondary Outcome: Maximum Flow Rate (Qmax)
Description: It's used to determine the degree of urinary difficulty.
Time Frame: 56 days
Population: For all subjects' medical histories in this study, there are one subject receiving Harnalidge 0.1 mg once daily (QD), 5 subjects receiving Harnalidge 0.2 mg QD, 22 subjects receiving Harnalidge 0.4 mg QD and eight subjects receiving Doxaben XL 4 mg QD for BPH treatment.
Measure: Mean (Standard Deviation); unit: ml/ sec
Arm/Group | Umooze | Placebo
Number analyzed (Participants) | 18 | 18
ml/ sec
  Qmax | 14.4 (4.29) | 12.72 (6.57)
  Difference of Qmax between V1 and V6 | 2.88 (3.77) | 2.49 (5.46)

3. Secondary Outcome: Postvoid Residual Volume (PVR)
Description: The PVR urine test measures the amount of urine left in the bladder after urination.
Time Frame: 56 days
Population: For all subjects' medical histories in this study, there are one subject receiving Harnalidge 0.1 mg once daily (QD), five subjects receiving Harnalidge 0.2 mg QD, 22 subjects receivingHarnalidge 0.4 mg QD and eight subjects receiving Doxaben 4 mg or Doxaben XL 4 mg QD for BPH treatment.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Umooze | Placebo
Number analyzed (Participants) | 18 | 18
ml
  Post- Void Residual Volume (PVR) | 35.3 (35.9) | 67.2 (47.8)
  Difference of PVR between V1 and V6 | -8.39 (31.9) | 14.8 (32.8)
Statistical Analysis 1: Comparison: Umooze vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

4. Secondary Outcome: Prostate Volume
Description: It's related to progression of benign prostatic hyperplasia (BPH).
Time Frame: 56 days
Population: For all subjects' medical histories in this study, there are one subject receiving Harnalidge 0.1 mg once daily (QD), five subjects receiving Harnalidge 0.2 mg QD, 22 subjects receiving Harnalidge 0.4 mg QD and eight subjects receiving Doxaben 4 mg or Doxaben XL 4 mg QD for BPH treatment.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Umooze | Placebo
Number analyzed (Participants) | 18 | 18
cm^3
  Prostate Volume | 29.1 (11.5) | 38.2 (20.1)
  Difference of prostate volume between V1 and V6 | -8.17 (12.7) | -1.33 (7.36)
Statistical Analysis 1: Comparison: Umooze vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

5. Secondary Outcome: Prostate-specific Antigen (PSA) Level
Description: Serum PSA test measures the amount of prostate- specific antigen in the blood. As a man's prostate enlarges with age, the amount of PSA in the blood normally increases.
Time Frame: 56 days
Population: For all subjects' medical histories in this study, there are one subject receiving Harnalidge 0.1 mg once daily (QD), five subjects receiving Harnalidge 0.2 mg QD, 22 subjects receiving 0.4 mg QD and eight subjects receiving Doxaben 4 mg or Doxaben XL 4 mg QD for BPH treatment.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Umooze | Placebo
Number analyzed (Participants) | 18 | 18
ng/ml
  Prostate- specific Antigen (PSA) | 1.67 (1.34) | 2.22 (1.69)
  Difference of PSA between V1 and V6 | 0.14 (0.32) | 0.26 (0.76)

6. Primary Outcome: Quality- Of- Life Index (QoL)
Description: The QoL index is a single question with scores of 0~6 point and corresponding to the assessment index ranging from delighted to terrible.
Time Frame: 56 days
Population: For all subjects' medical histories in this study, there are one subject receiving Harnalidge 0.1 mg once daily (QD), 5 subjects receiving Hatnalidge 0.2 mg QD, 22 subjects receiving Harnalidge 0.4 mg QD and eight subjects receiving Doxaben XL 4 mg QD for BPH treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Umooze | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  Quality-of-Life (QoL) | 2.72 (1.07) | 3.22 (1.17)
  Difference of QoL between V1 and V6 | -0.61 (1.20) | -0.56 (1.20)

7. Primary Outcome: International Prostate Symptom Score (IPSS) Between V1 and V6 in the Same Medication for More Than 12 Months
Description: as for outcome 1
Time Frame: 56 days
Population: All these five subjects in this statistical result have been treated BPH with 0.4 mg of Harnalidge for more than 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Umooze: Tablet oral dosage. Astragalus radix Extracts 480 mg+ Soy bean Extracts 20 mg
  Umooze: Umooze is consisted of Astragalus radix extracts and soy isoflavones. Astragalus radix (AR) is the dried root of Astragalus membranaceus Bge. Var. mongholicus and is used as a tonic in the traditional Chinese medicine. According to the reports submitted by the National Cancer institute of American, people who eat soybean products can reduce the incidence rate for prostate cancer. The composition of Umooze is invented by Golden Biotechnology Corp. against prostatic hyperplasia. The study product is given as add- on therapy in BPH. All the eligible subjects included in this study have the history for benign prostate hyperplasia (BPH) and receive the medication for this condition. Each subject receives the study product in the morning and evening for a continuous 56- day. Each oral dose of Umooze was given 2 tablets with about 240 ml of water.
Arm/Group | Umooze | Placebo
Number analyzed (Participants) | 2 | 3
units on a scale
  International prostate symptom score | 11.00 (4.24) | 14.33 (3.21)
  Difference in IPSS between V1 and V6 | -9.50 (3.54) | -4.33 (1.53)
Statistical Analysis 1: Comparison: Umooze vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

8. Primary Outcome: Quality of Life (QoL) Index Between V1 and V6 for the Subjects Taking 0.4 mg Harnalidge
Description: The Quality of Life (QoL) is a single question with scores of 0~6 point and corresponding to the assessment index ranging from delighted to terrible.
Time Frame: 56 days
Population: All these twenty-two subjects included in this statistical result have been received 0.4 mg Harnalidge for BPH treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Umooze: Tablet oral dosage. Astragalus radix Extracts 480 mg+ Soy bean Extracts 20 mg
  Umooze: Umooze is consisted of Astragalus radix extracts and soy isoflavones. Astragalus radix (AR) is the dried root of Astragalus membranaceus Bge. Var. mongholicus and is used as a tonic in the traditional Chinese medicine. According to the reports submitted by the National Cancer institute of American, people who eat soybean products can reduce the incidence rate for prostate cancer. The composition of Umooze is invented by Golden Biotechnology Corp. against prostatic hyperplasia. The study product is given as add- on therapy in BPH. All the eligible subjects included in this study have the history for benign prostate hyperplasia (BPH) and receive the medication for this condition. Each subject receives the study product in the morning and evening for a continuous 56- day. Each oral dose of the study product was given 2 tablets with about 240 ml of water.
Arm/Group | Umooze | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale
  Quality of Life (QoL) | 2.73 (1.10) | 3.27 (1.10)
  Difference of QoL between V1 and V6 | -0.82 (0.87) | -0.09 (0.70)
Statistical Analysis 1: Comparison: Umooze vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 56 days
Groups:
- Umooze: Tablet oral dosage. Astragalus radix Extracts 480 mg+ Soy extract 20 mg
  Umooze: Umooze is consisted of Astragalus radix extracts and soy isoflavones. Astragalus radix (AR) is the dried root of Astragalus membranaceus Bge. Var. mongholicus and is used as a tonic in the traditional Chinese medicine. According to the reports submitted by the National Cancer institute of American, people who eat soybean products can reduce the incidence rate for prostate cancer. The composition of Umooze is invented by Golden Biotechnology Corp. against prostatic hyperplasia. Umooze is used as add- on therapy for the subjects who take the medication for benign prostate hyperplasia (BPH). Each subject receives the study product in the morning and evening for a continuous 56- day. Each oral dose of Umooze was given 2 tablets with about 240 ml of water.
Arm/Group | Umooze | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 2/20 | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umooze (N=20) | Placebo (N=21)
Insomnia (Nervous system disorders) | 0 (0) | 1 (2) — Insomnia happened to only one subject who has been withdrawn from this study.
Rush (Immune system disorders) | 2 (2) | 1 (2) — This event took place in both umooze and placebo groups, one subject in placebo group and two subjects in umooze group. Rush on these three affected subjects was mild. There was one subject of them was withdrawn from the placebo group.
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) — It happened to only one subject in the placebo group. This subject got it mild and has been withdrawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other